CLINICAL TRIAL: NCT04250064
Title: A Study of Low Dose Bevacizumab With Conventional Radiotherapy Alone in Diffuse Intrinsic Pontine Glioma
Acronym: LoBULarDIPG
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3201
Record Dates: First submitted 2020-01-07; First posted 2020-01-31 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: DIPG
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concurrent low-dose Bevacizumab (Experimental): Low-dose concurrent Bevacizumab with standard radiotherapy
  Interventions: Drug: Bevacizumab Injection
- Ultra-low-dose RT (Experimental): Ultra-low-dose RT
  Interventions: Radiation: Ultra-low-dose RT

INTERVENTIONS:
Drug: Bevacizumab Injection — Additional concurrent low-dose Bevacizumab with standard EBRT
  Other Names: Concurrent low-dose Bevacizumab
  Arms: Concurrent low-dose Bevacizumab
Radiation: Ultra-low-dose RT — Ultra-low-dose EBRT instead of standard dose RT
  Arms: Ultra-low-dose RT

SUMMARY:
In this study, the investigators are testing improvement in survival outcomes in DIPG patients when stratified with MR perfusion score and treated with the said protocol. Newly diagnosed DIPG patients will undergo MRI perfusion study in addition to the usual MRI at diagnosis and will be stratified into hyperperfused or hypoperfused tumours.

The hyperperfused patients will receive additional low dose Bevacizumab weekly with conventional standard radiotherapy.

The hypo-perfused patients will receive ultra-low-dose radiotherapy fractionation equivalent to conventional RT biological dose.

DETAILED DESCRIPTION:
In tumours like Diffuse pontine glioma (DIPG), the diagnosis itself spells a death sentence for the child affected. The current standard treatment is conventionally fractionated daily radiation treatment for 6 weeks which benefits 80-90% patients with temporary improvement in neurological function which gives survival up to 8-10 months. With research over several decades, none of the altered fractionation radiotherapy or additional chemotherapy or targeted agents has shown a significant difference in outcomes.

The investigators propose to do an MRI perfusion study in addition to usual MRI at diagnosis and stratify them into hyperperfused or hypoperfused based on the criteria from the investigator's previously published institutional experience in DIPG. The hyperperfused patients will receive additional low dose a drug called Bevacizumab weekly with conventional standard radiotherapy. It is hypothesized that low dose Bevacizumab will decrease hypoxia and improve the efficacy of conventional radiotherapy and in turn improve outcomes.

The hypo-perfused patients will receive ultra-low-dose radiotherapy fractionation equivalent to conventional RT biological dose. As it is assumed that hypoperfused tumours are radioresistant, the investigator hypothesis that the ultra-low dose radiotherapy may overcome that radioresistance as seen in GBM adult patients and may improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Tumour Diagnosis: Newly diagnosed non-disseminated treatment naïve DIPG by classic clinical AND radiographic finding.
2. Age: Patient must be 3 to 18 years of age at the time of diagnosis.
3. Performance Score: KPS > 12 y/o >/= 50 or LPS for < 12y >/= 50 assessed at enrollment.
4. Participants must have normal organ and marrow function as defined below within two weeks prior to enrollment:

   1. Hematological: Absolute neutrophil count > 1,000/mcL, Platelets> 100,000/mcL (transfusion independent), HB > 8gm/dL (can be transfused)
   2. Hepatic: Total bilirubin < 1.5 times the upper limit of normal; alanine aminotransferase [SGPT (ALT)] and aspartate aminotransferase [SGOT (AST)] < 5 times the institutional upper limit of normal.
   3. Renal: Serum creatinine which is less than 1.5x the upper limit of institutional normal for age or Glomerular Filtration Rate (GFR) > 70 ml/min/1.73m2.; The absence of clinically significant proteinuria as defined by a screening early morning urine (first sample) dipstick urinalysis of < 2.
   4. Normal coagulation profile
5. Post-Biopsy patients allowed, but should not have evidence of haemorrhage greater than 0.5cm intracranially and should satisfy this criterion within two to four weeks of biopsy to start treatment in Arm 1 if designated as per perfusion study along with satisfying other criteria as applicable. For arm 2, there will be no restriction other than the usual criteria.
6. No contra-indication for GA for MRI
7. Would not need GA for RT in the hypofractionated subgroup (due to logistics).
8. Ability to understand and the willingness to sign a written informed consent document by the parent or guardian and assent by the child as applicable and as per institutional policy.

Exclusion Criteria:

Other than those mentioned above,

1. Surgical Procedures: Patients who have had major surgery should not receive the first dose of BVZ until 28 days after major surgery or Serious or Non-Healing Wounds
2. Patients with uncontrolled systemic hypertension/ Proteinuria with a urine protein (albumin)/creatinine ratio of ≥1.0.
3. Thrombosis: Patients must not have been previously diagnosed with a deep venous or arterial thrombosis (including pulmonary embolism), and must not have a known thrombophilic condition.
4. Allergies: Patients with a history of allergic reaction to Chinese hamster ovary cell products, or other recombinant human antibodies.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | median of 12 months from diagnosis
  Survival for the total enrolled patient population will calculated at the median follow up 12 months. This will be compared with historical data from TMH, international DIPG registry and SIOP DIPG registry for 12-month OS as 35%.

SECONDARY OUTCOMES:
Progression-free survival | 6 months, 12 months, 18 months from diagnosis
  Progression-free survival: at 6 months, 12 months, 18 months will be recorded for overall cohort and each arm separately at first progression only. For the purpose of the study, any patient with two or more new clinical signs of neurological deterioration in accordance with classical DIPG diagnosis with radiological progression of disease from any previous available imaging will be called progression.
Adverse events | From the time of intervention beginning, through the course of intervention, at the end of intervention and follow up 3 monthly to the date of precluding progression, or last known follow-up date, assessed for up to 2 years
  The documentation of highest grade of toxicity as per CTCAE v 4 and RTOG radiation toxicity.
Steroid Use | From the time of intervention beginning, through the course of intervention, at the end of intervention and follow up 3 monthly to the date of precluding progression, or last known follow-up date, assessed for up to 2 years
  Total duration of steroid use will be recorded
Pattern of relapse | from the date of enrollment on study to the last known follow-up date, assessed for up to 2 years
  local versus disseminated progression will be documented for each arm and overall cohort for the patients with available MRI at progression.
Overall survival | 6, 12 month and 18 months.
  Overall survival in each arm as well as for overall cohort will be recorded
Compliance | From the time of intervention beginning, through the course of intervention, till the planned intervention is completed to maximum of 10 weeks from beginning , which ever is earlier.
  Treatment intervention abandonment rates: number of patients not completing the planned intervention/treatment.
Inconvenience rates | From the time of intervention beginning, through the course of intervention, till the end of intervention or maximum of upto 10 weeks, which ever is earlier.
  average number of hours spent in hospital per day during the intervention phase.
Quality of Life scores | From date of accrual until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  The Qol scores will be calculated as per the routine OPD based collection of Health using utilities index (40 item standard questionnaire) and/or PedQol interviewer based scores.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Krishnatry, Dr, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India